CLINICAL TRIAL: NCT04798092
Title: Impact of Parathyroidectomy on Renal Function in Patients With Primary Hyperparathyroidism
Brief Title: Impact of Parathyroidectomy on Renal Function
Acronym: PARA-REIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI099
Record Dates: First submitted 2021-01-29; First posted 2021-03-15 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-01

CONDITIONS: Primary Hyperparathyroidism
Keywords: Primary Hyperparathyroidism; Renal function
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Parathyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: parathyroidectomy — surgical removal of parathyroid adenoma(s) with postoperative biological cure

SUMMARY:
Primary hyperparathyroidism (PHPT) is a disorder of one or more of the parathyroid glands. The parathyroid gland(s) becomes overactive and secretes excess amounts of parathyroid hormone (PTH). As a result, the blood calcium rises to a level that is higher than normal. PHPT is associated with several other metabolic complications as osteoporosis, kidney stones, hypertension, insulin resistance, cardiac calcifications, cardiac arrhythmias, and kidney failure. Renal function deterioration over time has also been reported. However, the role of parathyroidectomy on renal function remains controversial in patients with PHPT. In some studies, surgical cure of PHPT has been shown to halt renal function deterioration in patients with coexisting renal disease. On the other hand, other studies showed no significant impact of parathyroidectomy on renal function. Consequently, the goal of this study was to evaluate renal function before and after parathyroidectomy in a large cohort of patients with pHPT.

DETAILED DESCRIPTION:
Primary hyperparathyroidism (PHPT) is a disorder of one or more of the parathyroid glands. The parathyroid gland(s) becomes overactive and secretes excess amounts of parathyroid hormone (PTH). As a result, the blood calcium rises to a level that is higher than normal. PHPT is associated with several other metabolic complications as osteoporosis, kidney stones, hypertension, insulin resistance, cardiac calcifications, cardiac arrhythmias, and kidney failure. Renal function deterioration over time has also been reported. However, the role of parathyroidectomy on renal function remains controversial in patients with PHPT. In some studies, surgical cure of PHPT has been shown to halt renal function deterioration in patients with coexisting renal disease. On the other hand, other studies showed no significant impact of parathyroidectomy on renal function. Consequently, the goal of this study was to evaluate renal function before and after parathyroidectomy in a large cohort of patients with pHPT.

Criteria are detailled in "Outcomes measures"

ELIGIBILITY:
Inclusion Criteria:

- patients undergoing parathyroidectomy for primary hyperparathyroidism with surgical cure defined as postoperative normocalciemia

Exclusion Criteria:

* patients on dialysis
* GFR < 15 ml/min
* renal graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing parathyroidectomy for primary hyperparathyroidism with surgical cure defined as postoperative normocalciemia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change in renal function | preoperative, postoperative at 3, 6, and 12 months
  glomerular filtration rate (CKD in mL/min)

SECONDARY OUTCOMES:
Change in calcium | preoperative, postoperative at 3, 6, and 12 months
  Blood calcium level (in mg/L)
Change in parathormone | preoperative, postoperative at 3, 6, and 12 months
  Blood parathormone level (in ng/dL)
Change in vitamin D | preoperative, postoperative at 3, 6, and 12 months
  Blood vitamine D level (in ng/mL)
Change in urinary calcium | preoperative, postoperative at 3, 6, and 12 months
  Urine calcium level (in mg/24h)
Change in insulin | preoperative, postoperative at 3, 6, and 12 months
  Fasting blood insuline level (in mUI/L)
Change in glycemia | preoperative, postoperative at 3, 6, and 12 months
  Fasting blood glucose level (in g/L)
Change in osteocalcin | preoperative, postoperative at 3, 6, and 12 months
  Blood osteocalcin level (in ng/mL)
Change in bone alkaline phosphatases | preoperative, postoperative at 3, 6, and 12 months
  Blood bone alkaline phosphatases level (in microgr/L)
Change in aldosterone | preoperative, postoperative at 3, 6, and 12 months
  Blood aldosterone level (in pg/mL)
Change in renin | preoperative, postoperative at 3, 6, and 12 months
  Blood active renin (in pg/mL)
Change in total cholesterol | preoperative, postoperative at 3, 6, and 12 months
  Blood total cholesterol (in gr/L)
Change in HDL cholesterol | preoperative, postoperative at 3, 6, and 12 months
  Blood HDL Cholesterol (in gr/L)
Change in LDL cholesterol | preoperative, postoperative at 3, 6, and 12 months
  Blood LDL Cholesterol (in gr/L)
Change in triglycerides | preoperative, postoperative at 3, 6, and 12 months
  Blood triglycerides (in gr/L)
CAC scoring on CT scan | preoperative
  CAC score (actual value)

CONTACTS AND LOCATIONS:
Overall Officials: Brunaud, Principal Investigator — CHU NANCY
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided